CLINICAL TRIAL: NCT02378207
Title: A Randomized, Placebo-controlled, Partially Blinded Phase 1b Clinical Trial to Evaluate the Safety and Immunogenicity of BCG Revaccination, H4:IC31, and H56:IC31 in Healthy, HIV-1-Uninfected Adolescent Participants
Brief Title: Safety and Immunogenicity Study of BCG, H4:IC31, and H56:IC31 Revaccination in Healthy Adolescents
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Aeras (Other)
Collaborators: HIV Vaccine Trials Network (Network); Sanofi Pasteur, a Sanofi Company (Industry); Statens Serum Institut (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: HVTN 602 / AERAS A-042
Record Dates: First submitted 2015-02-12; First posted 2015-03-04 (Estimated); Results first posted 2019-11-18 (Actual); Last update posted 2019-11-18 (Actual); Status verified 2018-01

CONDITIONS: Tuberculosis
MeSH Terms: conditions — Tuberculosis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Group 1 H4:IC31 (Experimental): 15 mcg H4/500 nmol IC31 administered IM as 0.5 mL in alternating deltoid muscle at Days 0 and 56.
  Interventions: Biological: H4:IC31
- Group 2 H56:IC31 (Experimental): 5 mcg H56/500 nmol IC31 administered IM as 0.5 mL in alternating deltoid muscle at Days 0 and 56.
  Interventions: Biological: H56:IC31
- Group 3 BCG (2-8 x 105 CFU) (Active Comparator): Administered IM as 0.1 mL in either deltoid muscle at Day 0.
  Interventions: Biological: BCG
- Group 4 Control Sodium Chloride 0.9% (Placebo Comparator): Administered IM as 0.5 mL in alternating deltoid muscle at Days 0 and 56.
  Interventions: Biological: Control Sodium Chloride 0.9%

INTERVENTIONS:
Biological: H4:IC31 — H4 contains Mtb antigens Ag85B and TB10.4
  Arms: Group 1 H4:IC31
Biological: H56:IC31 — H56 contains Mtb antigens ESAT-6, and Rv2660c
  Arms: Group 2 H56:IC31
Biological: BCG
  Arms: Group 3 BCG (2-8 x 105 CFU)
Biological: Control Sodium Chloride 0.9%
  Arms: Group 4 Control Sodium Chloride 0.9%

SUMMARY:
The aims of the phase 1b trial described here are to facilitate identification of assays and immune responses that could then be evaluated as correlates of risk and correlates of protection in efficacy studies and ultimately to provide leads for biomarkers of protection against tuberculosis. This study will complement one ongoing study (NCT02075203) evaluating the prevention of M. Tuberculosis infection using H4:IC31 (also known as AERAS-404).

DETAILED DESCRIPTION:
This study proposes to further evaluate the safety and immunogenicity of H4:IC31, H56:IC31, and BCG revaccination. The study will be conducted in previously BCG vaccinated healthy adolescents, and will entail a thorough immunogenicity evaluation of these regimens incorporating unbiased systems vaccinology approaches and novel assessments of baseline and elicited responses that may impact vaccine responses. A major goal for this study is to generate immunological data on a wide range of immune responses using a variety of approaches including validated assessments, unbiased strategies, and novel exploratory assays to increase the likelihood of detecting responses correlating with risk or protection in the prevention of infection study. Investigators contributing to the proposed study have participated in a correlates analysis for an HIV vaccine exhibiting modest efficacy in which 2 correlates of risk were identified.

An additional aim of this study is to explore factors affecting vaccine induced responses that may also impact efficacy. For example, it is hypothesized that exposure to environmental mycobacteria may alter protection provided by BCG vaccination. Reagents for evaluating levels of exposure to environmental mycobacteria are in development as part of a concurrent collaborative study. An exploratory objective for this trial is to apply these reagents to examine whether such exposures influence immune responses elicited by the study vaccine and regimens.

ELIGIBILITY:
Inclusion Criteria:

1. Age of 12 to ≤ 17 years at enrollment
2. Minimum weight ≥ 40 kg
3. Previous BCG vaccination at least 5 years ago documented by scarification or medical card
4. No evidence of active TB disease, as determined by history, physical examination and, if deemed appropriate, sputum investigation and / or chest x-ray.
5. Negative QFT-GIT test at screening, using the manufacturer's recommended threshold of 0.35 IU/mL
6. Assessed by the clinic staff as being at low risk for HIV infection
7. Hemoglobin ≥ 11.7 g/dL for females, ≥ 12.5 g/dL for males
8. Negative HIV-1 and -2 blood test
9. Agree to consistently use effective contraception for sexual activity that could lead to pregnancy from at least 20 days prior to enrollment through the last required protocol clinic visit.

(additional minor criteria not added due to space constraints)

Exclusion Criteria:

1. Blood products received within 120 days before first vaccination
2. Investigational research agents received within 182 days before first vaccination
3. Intent to participate in another study of an investigational research agent during the planned duration of the HVTN 602 / AERAS A-042 study
4. Pregnant or breastfeeding
5. History of alcohol or drug abuse
6. A significant contact with active TB disease: for example, shared residency with an individual receiving anti-TB treatment, or with an individual known to have incompletely treated culture or smear positive TB
7. TB prophylaxis within 90 days prior to enrollment
8. History of treatment for active TB disease or latent Mtb infection
9. Positive and indeterminate QFT-GIT result
10. Received a tuberculin skin test (TST) within 90 days prior to enrollment
11. Vaccines and other Injections
12. Immunosuppressive medications received within 168 days before first vaccination.
13. Serious adverse reactions to vaccines including history of anaphylaxis and related symptoms such as hives, respiratory difficulty, angioedema, and/or abdominal pain.
14. Immunoglobulin received within 60 days before first vaccination
15. Autoimmune disease Not excluded: mild, well-controlled psoriasis
16. Clinically significant medical condition, physical examination findings, clinically significant abnormal laboratory results, or past medical history with clinically significant implications for current health. Including but not limited to: Diabetes mellitus type 1 or type 2, Thyroidectomy, or Thyroid disease, Asthma, Asplenia, Bleeding disorders, malignancy, Seizure disorder, and Angioedema

(additional minor criteria not added due to space constraints)

Ages: 12 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 84 (Actual)
Dates: Start 2015-05; Primary Completion 2016-10-31 (Actual); Study Completion 2016-12-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Linda-Gail Bekker, MD, Study Chair — Desmond Tutu HIV Centre; Jim Kublin, MD, Study Chair — HVTN Core, FHCRC
Locations (1):
- Desmond Tutu HIV Foundation, Cape Town, South Africa

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Bekker LG, Dintwe O, Fiore-Gartland A, Middelkoop K, Hutter J, Williams A, Randhawa AK, Ruhwald M, Kromann I, Andersen PL, DiazGranados CA, Rutkowski KT, Tait D, Miner MD, Andersen-Nissen E, De Rosa SC, Seaton KE, Tomaras GD, McElrath MJ, Ginsberg A, Kublin JG; HVTN 602/Aeras A-042 Protocol Team. A phase 1b randomized study of the safety and immunological responses to vaccination with H4:IC31, H56:IC31, and BCG revaccination in Mycobacterium tuberculosis-uninfected adolescents in Cape Town, South Africa. EClinicalMedicine. 2020 Mar 18;21:100313. doi: 10.1016/j.eclinm.2020.100313. eCollection 2020 Apr. PMID 32382714

RESULTS

PARTICIPANT FLOW:
Groups:
- Group 3 BCG (2-8 x 105 CFU): Administered ID as 0.1 mL in either deltoid muscle at Day 0.
Period: Overall Study
Arm/Group | Group 1 H4:IC31 | Group 2 H56:IC31 | Group 3 BCG (2-8 x 105 CFU) | Group 4 Control Sodium Chloride 0.9%
Started | 24 | 24 | 24 | 12
Completed | 24 | 21 | 22 | 11
Not Completed | 0 | 3 | 2 | 1

BASELINE CHARACTERISTICS:
Groups:
- Group 1 H4:IC31: 15 mcg H4/500 nmol IC31 administered IM as 0.5 mL in alternating deltoid muscle at Days 0 and 56.
  n=24
- Group 2 H56:IC31: 5 mcg H56/500 nmol IC31 administered IM as 0.5 mL in alternating deltoid muscle at Days 0 and 56.
  n=24
- Group 3 BCG (2-8 x 105 CFU): Administered ID as 0.1 mL in either deltoid muscle at Day 0.
  n=24
- Group 4 Control Sodium Chloride 0.9%: Administered IM as 0.5 mL in alternating deltoid muscle at Days 0 and 56.
  n=24
- Total: Total of all reporting groups
Arm/Group | Group 1 H4:IC31 | Group 2 H56:IC31 | Group 3 BCG (2-8 x 105 CFU) | Group 4 Control Sodium Chloride 0.9% | Total
Number analyzed (Participants) | 24 | 24 | 24 | 12 | 84
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 24 | 24 | 24 | 12 | 84
  Between 18 and 65 years | 0 | 0 | 0 | 0 | 0
  >=65 years | 0 | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 13.8 (1.42) | 13.7 (1.46) | 14.5 (1.47) | 13.2 (1.11) | 13.9 (1.45)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 13 | 11 | 6 | 45
  Male | 9 | 11 | 13 | 6 | 39
Region of Enrollment [Number; unit: participants]
  South Africa | 24 | 24 | 24 | 12 | 84
Participants: QuantiFERON-TB Gold In-Tube (QFT-GIT)-negative, HIV-negative, and BCG vaccinated [Count of Participants; unit: Participants] | 24 | 24 | 24 | 12 | 84

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Adverse Events
Description: The number of solicited and unsolicited adverse events (AEs), including serious adverse events (SAEs), recorded post-vaccination for all participants.
Time Frame: Up to 8 months
Measure: Number; unit: participants
Arm/Group | Group 1 H4:IC31 | Group 2 H56:IC31 | Group 3 BCG (2-8 x 105 CFU) | Group 4 Control Sodium Chloride 0.9%
Number analyzed (Participants) | 24 | 24 | 24 | 12
participants | 22 | 20 | 24 | 10

2. Primary Outcome: Percentage of Participants With Response Rates to TB Antigens as Compared to Baseline
Description: Flow cytometry was used to examine TB Mb-specific CD4+ and CD8+ T-cell responses using the ICS assay. The antigens used to stimulate cells in this assay included peptide pools for the vaccine-matched proteins (Ag85B, ESAT-6, Rv2660c, and TB 10.4) as well as complex TB antigens (TB whole cell lysate [TB WCL], and BCG Pasteur strain.
Time Frame: Days 70 and 168
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Group 1 H4:IC31 | Group 2 H56:IC31 | Group 3 BCG (2-8 x 105 CFU) | Group 4 Control Sodium Chloride 0.9%
Number analyzed (Participants) | 24 | 24 | 24 | 12
percentage of participants
  Response rates to Ag85B on Day 70 | 40.0 [21.9 to 61.3] | 45.0 [25.8 to 65.8] | 0.0 [0.0 to 17.6] | 0.0 [0.0 to 25.95]
  Response rates to TB10.4 on Day 70 | 21.1 [8.5 to 43.3] | 5.6 [1.0 to 25.8] | 5.9 [1.0 to 27.0] | 0.0 [0.0 to 25.9]
  Response rates to Ag85B on Day 168 | 21.7 [9.7 to 41.9] | 9.5 [2.7 to 28.9] | 4.3 [0.8 to 21.0] | 0.0 [0.0 to 27.8]
  Response rate to TB10.4 on Day 168 | 8.7 [2.4 to 26.8] | 0.0 [0.0 to 15.5] | 0.0 [0.0 to 14.3] | 0.0 [0.0 to 27.8]

3. Secondary Outcome: Evaluate Humoral Responses Elicited by the Different Vaccine Regimens.
Description: Vaccine-specific binding antibodies elicited by the vaccine regimens as determined by multiplex antibody assay and/or enzyme-linked immunosorbent assay (ELISA).
Time Frame: Up to day 168.
Reporting Status: Not Posted

4. Secondary Outcome: * Evaluate Immune Response From Vaccine Regimens by Measuring Early (Innate) Vaccine-induced Peripheral Blood Transcription Profiles; Determine Which Responses Are Associated With Antigen-specific Adaptive Responses * Evaluate Adaptive Immune Response.
Description: * Changes in gene expression measured in longitudinally-collected blood samples relative to samples collected at baseline. The transcriptional profiles will be correlated with antigen-specific adaptive responses measured in Primary objective 2.
  * Transcriptional analysis of antigen-stimulated peripheral blood mononuclear cells (PBMC) at 2 weeks post vaccination will be performed..
Time Frame: Up to day 168
Reporting Status: Not Posted

5. Secondary Outcome: Evaluate Changes in Innate Cells in Response to the Vaccine Regimens
Description: Blood concentrations of innate immune cell populations including lymphocyte populations, dendritic cells, monocytes, and granulocytes before and after vaccination
Time Frame: Up to day 168
Reporting Status: Not Posted

6. Secondary Outcome: Measure Non-classical Major Histocompatibility Complex (MHC)-Restricted T-cell Vaccine-induced Responses, Such as to Mycobacterial Lipids (CD1-restricted) and Metabolites (MR1-restricted).
Description: * Frequency of CD4+, CD8+, and CD4/CD8 double-negative T-cell responses restricted by CD1 (recognizing specific Mtb lipids) before and after BCG revaccination in Group 3 participants.
  * Frequency of mucosal-associated invariant T-cells (MAIT) restricted by MR1 (recognizing vitamin B metabolites) before and after BCG revaccination in Group 3 participants
Time Frame: Up to day 168
Reporting Status: Not Posted

7. Secondary Outcome: Evaluate QFT-GIT and ESAT-6 Free IGRA Discordance and Conversion/Reversion Rate During the Course of the Trial.
Description: * Magnitude and positivity of interferon (IFN)-γ release using QFT-GIT ELISA in QFT-GIT tests.
  * Magnitude and positivity of IFN-γ release using QFT-GIT ELISA in ESAT-6 free IGRAs.
Time Frame: Up to day 168
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: AEs: 7 days post each vaccination Unsolicited AEs: 28 days post each vaccination Solicited injection-site reaction AEs: BCG group - 84 days post each vaccination; H4:IC31/placebo - 28 days post each vaccination; H56:IC31/placebo - 28 days post each vaccination SAEs, AEs of special interest, SUSARs: through day 224
Groups:
- Group 1 H4:IC31: 15 mcg H4/500 nmol IC31 administered IM as 0.5 mL in alternating deltoid muscle at Days 0 and 56.
  H4:IC31
- Group 2 H56:IC31: 5 mcg H56/500 nmol IC31 administered IM as 0.5 mL in alternating deltoid muscle at Days 0 and 56.
  H56:IC31
- Group 3 BCG (2-8 x 105 CFU): Administered ID as 0.1 mL in either deltoid muscle at Day 0.
  BCG
- Group 4 Control Sodium Chloride 0.9%: Administered IM as 0.5 mL in alternating deltoid muscle at Days 0 and 56.
  Control Sodium Chloride 0.9%
Arm/Group | Group 1 H4:IC31 | Group 2 H56:IC31 | Group 3 BCG (2-8 x 105 CFU) | Group 4 Control Sodium Chloride 0.9%
All-Cause Mortality (participants affected / at risk) | 0/24 | 0/24 | 0/24 | 0/12
Serious Adverse Events (participants affected / at risk) | 0/24 | 1/24 | 1/24 | 0/12
Other Adverse Events (participants affected / at risk) | 22/24 | 20/24 | 24/24 | 10/12
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group 1 H4:IC31 (N=24) | Group 2 H56:IC31 (N=24) | Group 3 BCG (2-8 x 105 CFU) (N=24) | Group 4 Control Sodium Chloride 0.9% (N=12)
Impetigo (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Road traffic accident (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cardiac murmur functional (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group 1 H4:IC31 (N=24) | Group 2 H56:IC31 (N=24) | Group 3 BCG (2-8 x 105 CFU) (N=24) | Group 4 Control Sodium Chloride 0.9% (N=12)
Palpitations (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (4)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Aphthous stomatitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 1 (3) | 6 (6) | 2 (2)
Nausea (Gastrointestinal disorders) | 3 (3) | 5 (7) | 3 (3) | 1 (1)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Chills (General disorders) | 5 (7) | 6 (7) | 2 (3) | 2 (3)
Fatigue (General disorders) | 6 (10) | 7 (12) | 8 (9) | 1 (1)
Feeling cold (General disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Implant site swelling (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Injection site erythema (General disorders) | 2 (3) | 4 (6) | 0 (0) | 0 (0)
Injection site pain (General disorders) | 14 (16) | 13 (21) | 0 (0) | 3 (6)
Injection site pruritus (General disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Injection site swelling (General disorders) | 3 (4) | 4 (4) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 2 (2) | 2 (2) | 0 (0) | 1 (1)
Vaccination site discolouration (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Vaccination site erythema (General disorders) | 0 (0) | 0 (0) | 8 (8) | 0 (0)
Vaccination site exfoliation (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Vaccination site induration (General disorders) | 0 (0) | 0 (0) | 10 (10) | 0 (0)
Vaccination site pain (General disorders) | 0 (0) | 0 (0) | 14 (18) | 0 (0)
Vaccination site pruritus (General disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Vaccination site rash (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Vaccination site scab (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Vaccination site scar (General disorders) | 0 (0) | 0 (0) | 3 (3) | 0 (0)
Vaccination site swelling (General disorders) | 0 (0) | 0 (0) | 13 (13) | 0 (0)
Vaccination site ulcer (General disorders) | 0 (0) | 0 (0) | 7 (7) | 0 (0)
Cellulitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Folliculitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gastroenteritis viral (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Influenza (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Lower respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pharyngitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Rhinitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Trichomoniasis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Vaccination site abscess (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Viral upper respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Blood pressure diastolic increased (Investigations) | 5 (7) | 2 (5) | 4 (4) | 1 (1)
Blood pressure systolic increased (Investigations) | 4 (4) | 5 (7) | 4 (4) | 2 (2)
Neutrophil count decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Protein urine (Investigations) | 5 (6) | 1 (1) | 2 (2) | 2 (2)
White blood cell count increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 3 (5) | 3 (4) | 1 (2)
Myalgia (Musculoskeletal and connective tissue disorders) | 2 (2) | 5 (6) | 4 (4) | 1 (1)
Dizziness (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 7 (9) | 6 (8) | 8 (8) | 2 (2)
Haemorrhage in pregnancy (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Haematuria (Renal and urinary disorders) | 2 (2) | 3 (3) | 0 (0) | 0 (0)
Proteinuria (Renal and urinary disorders) | 3 (3) | 2 (3) | 1 (1) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Rash papular (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No